CLINICAL TRIAL: NCT00073385
Title: A Randomized Trial of Pivanex Plus Docetaxel or Docetaxel Monotherapy in Patients With Chemotherapy Resistant Advanced Non-Small Cell Carcinoma of the Lung (NSCLC)
Brief Title: Comparative Trial of Pivanex and Docetaxel Vs Docetaxel Monotherapy in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Titan Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTP-200-03-01; NSCLC Clincal Trial
Record Dates: First submitted 2003-11-19; First posted 2003-11-21 (Estimated); Last update posted 2005-08-30 (Estimated); Status verified 2005-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung cancer, Docetaxel, Histone deacetylase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pivalyloxymethyl butyrate; Docetaxel

INTERVENTIONS:
Drug: Pivanex
Drug: Docetaxel

SUMMARY:
This randomized study will assess the efficacy and safety of the combination of Pivanex and docetaxel compared to docetaxel alone in patients with a type of lung cancer called non-small cell lung cancer. Pivanex is an investigational agent, and docetaxel is an approved drug.

DETAILED DESCRIPTION:
Rationale: Pivanex is a histone deacetylase inhibitor that induces tumor differentiation and/or apoptosis. Pivanex has been well tolerated in clinical trials and has shown preliminary evidence of efficacy in patients with non-small cell lung cancer. Docetaxel is an approved drug for second-line treatment of non-small cell lung cancer. Preclinical studies indicate that the combination of Pivanex and docetaxel is synergistic.

Purpose: This open-label randomized trial will evaluate whether combination therapy with Pivanex and docetaxel provides clinical benefit over docetaxel alone in patients with chemotherapy resistant non-small cell lung cancer.

Objectives:

* Compare the survival of patients with non-small cell lung cancer treated with combination therapy with Pivanex and docetaxel vs. docetaxel alone
* Compare the time to disease progression, tumor responses, and safety profile of patients with non-small cell lung cancer treated with combination therapy with Pivanex and docetaxel vs. docetaxel alone

Outline: This is a randomized, open-label, multicenter study in patients with non-small cell lung cancer who have previously been treated with no more than one prior platinum containing chemotherapy regimen. Patients are stratified by ECOG performance status (0-1 vs. 2), response to prior platinum based chemotherapy (progression vs. CR/PR/SD) and prior taxane therapy (yes vs. no). Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive the combination of Pivanex intravenously on Days 1-3 and docetaxel intravenously on Day 4. Treatment repeats every 21 days until disease progression or treatment withdrawal.
* Arm B: Patients receive docetaxel intravenously on Day 1. Treatment repeats every 21 days until disease progression or treatment withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC); Treatment with one prior platinum-based chemotherapy regimen (Eligible patients may include:

  1. Patients previously treated with adjuvant or neoadjuvant chemotherapy (must be completed within 6 months prior to randomization) or
  2. Patients who have received chemotherapy for advanced or metastatic lung cancer);
* Recurrent or progressive NSCLC (local, distant, or both) following initial chemotherapy);
* Measurable or non-measurable disease;
* Males and females, age => 18 years;
* Adequate renal function with creatinine => 1.5 mg/dl;
* Adequate liver function with alkaline phosphatase => 2.5 X upper limit of normal, SGOT, and SGPT => 1.5 X upper limit of normal; and total bilirubin => upper limit of normal;
* Adequate bone marrow function: platelets > 100,000/mm3, hemoglobin => 9 g/dL, and absolute neutrophil count (ANC) => 1,500 cells/mm3;
* Able to give informed consent;
* Discontinuation of previous surgery, radiation therapy or cancer chemotherapy at least four weeks prior to randomization (six weeks if a prior nitrosourea or mitomycin C), with recovery from treatment-associated toxicity;
* A predicted life expectancy of at least 12 weeks; and
* ECOG performance status of 0, 1, or 2.

Exclusion Criteria:

* Receipt of more than one chemotherapy regimen for NSCLC;
* A second malignancy within the last 5 years other than curatively treated carcinoma-in-situ or non-melanoma skin cancer;
* Pregnant or lactating females (Females of childbearing potential must have a negative pregnancy test and all male and female patients of reproductive potential must agree to use adequate birth control);
* Known HIV-positive patients;
* Acute medical problems, such as ischemic heart or lung disease or uncontrolled systemic infection;
* Patients with any underlying medical conditions or circumstance, which would contraindicate therapy with study treatment, affect compliance or impair evaluation of study endpoints;
* Patients receiving investigational agents within 30 days of the screening visit;
* Known allergy to reagents in the study;
* Prior docetaxel therapy;
* Symptomatic or untreated brain metastases (Patients with brain metastases are eligible if they are clinically and neurologically stable for > 4 weeks since therapy (radiation therapy, radiosurgery/gamma knife; surgical resection) as determined by the investigator and either off corticosteroids or on a stable dose of corticosteroids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225
Dates: Start 2003-09; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Wilshire Oncology Medical Group, La Verne, California
  - Hematology and Oncology Specialists, LLC, New Orleans, Louisiana
  - HemOnCare, Brooklyn, New York
  - Montefiore Medical Center, Department of Oncology, The Bronx, New York
  - Gaston Hematology & Oncology Associates, Gastonia, North Carolina
- India (2):
  - Rajiv Gandhi Cancer Institute & Research Center, New Delhi
  - Regional Cancer Centre, Thiruvananthapuram
- University of Edinburgh, Edinburgh Cancer Centre, Edinburgh, United Kingdom